CLINICAL TRIAL: NCT05977322
Title: A Phase I, Open-label, Multi-center Study to Evaluate the Safety, Tolerability, Dosimetry and Preliminary Activity of [177Lu]Lu-FF58 in Patients With Selected Advanced Solid Tumors.
Brief Title: A Phase I Study of [177Lu]Lu-FF58 in Patients With Advanced Solid Tumors.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision was not based on any safety concerns
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAA604A12101; 2020-502367-37-00 (Other: EU CTIS)
Record Dates: First submitted 2023-07-10; First posted 2023-08-04 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Gastroesophageal Adenocarcinoma; Glioblastoma Multiforme
Keywords: pancreatic ductal adenocarcinoma; PDAC; pancreatic cancer; gastroesophageal adenocarcinoma; GEA; gastric cancer; gastric adenocarcinoma; esophageal cancer; esophageal adenocarcinoma; glioblastoma multiforme; GBM; advanced solid tumors; radioligand therapy; RLT; [177Lu]Lu-FF58; [68Ga]Ga-FF58; integrins; alpha-v beta-3 integrin; αvβ3; alpha-v beta-5 integrin; αvβ5
MeSH Terms: conditions — Glioblastoma; Pancreatic Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Patients will receive 68Ga-FF58 and only patients with tumor uptake of 68Ga-FF58 will receive 177Lu-FF58.
  Interventions: Drug: 68Ga-FF58; Drug: 177Lu-FF58

INTERVENTIONS:
Drug: 68Ga-FF58 — Kit for radiopharmaceutical preparation of 68Ga- FF58 solution for injection
Drug: 177Lu-FF58 — Solution for injection/infusion

SUMMARY:
The purpose of the study is to test the safety and dosing of [177Lu]Lu-FF58, a radioligand therapy for patients with advanced or metastatic tumors that express proteins known as integrins: alpha-v beta-3 integrin (αvβ3) and alpha-v beta-5 integrin (αvβ5). The study will also further characterize the radioligand imaging agent [68Ga]Ga-FF58 including its ability to identify tumor lesions and its safety profile.

DETAILED DESCRIPTION:
The study will be done in two parts. The first part is called "escalation" and the second part is called "expansion". In both parts of the study, patients will be screened with a [68Ga]Ga-FF58 positron emission tomography (PET)/computed tomography (CT) or PET/magnetic resonance imaging (MRI) scan to assess eligibility for treatment with [177Lu]Lu-FF58. In the escalation part, different doses of [177Lu]Lu-FF58 will be tested to identify the recommended dose. The expansion part of the study will examine the safety and preliminary efficacy of [177Lu]Lu-FF58 at the recommended dose determined during the escalation part. The end of study will occur when at least 80% of the patients in the expansion part have completed the follow-up for disease progression or discontinued from the study for any reason, and all patients have completed treatment and the 36 month long term follow- up period, or the study is terminated early in which case all patients would also be followed up for safety.

ELIGIBILITY:
Key Inclusion criteria

* Age >= 18 years old
* Patients with locally advanced unresectable or metastatic PDAC, locally advanced unresectable or metastatic GEA, or recurrent GBM
* To be treated with [177Lu]Lu-FF58, patients must have at least one measurable lesion that shows [68Ga]Ga-FF58 uptake on PET/CT or PET/MRI

Key Exclusion criteria

* Absolute neutrophil count (ANC) < 1.5 x 109/L, hemoglobin < 10 g/dL, or platelet count < 100 x 109/L
* Prior external beam radiation therapy (EBRT) to > 25% of the bone marrow
* Creatinine clearance < 60 mL/min
* Unmanageable bladder outflow obstruction or urinary incontinence
* Non-GBM patients: Presence of symptomatic central nervous system (CNS) metastases, or CNS metastases that require local CNS-directed therapy (such as radiotherapy or surgery), or increasing doses of corticosteroids within 1 week before [177Lu]Lu-FF58 administration

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of dose limiting toxicities of 177Lu-FF58 | From start of study treatment until 6 weeks after
  A dose limiting toxicity (DLT) is defined as any AE or abnormal laboratory value of CTCAE (v5.0) Grade 3 or higher that occurs within the DLT evaluation period (i.e., 6 weeks starting from the first administration of 177Lu-FF58) and that is not primarily related to disease, disease progression, intercurrent illness, or concomitant medications.
Incidence and severity of adverse events and serious adverse events of 177Lu-FF58 | From start of study treatment until 180 days after the last dose of study treatment, assessed up to approximately 15 months
  The distribution of adverse events will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs) and Serious Adverse Event (TESAEs) due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.
Dose modifications for 177Lu-FF58 | From start of study treatment until last dose of study treatment, assessed up to approximately 36 weeks
  Dose modifications (dose interruptions and reductions) for 177Lu-FF58 will be assessed and summarized using descriptive statistics. The number of patients with dose modification and the reasons will be summarized by treatment groups.
Dose intensity for 177Lu-FF58 | From start of study treatment until last dose of study treatment, assessed up to approximately 36 weeks
  Dose intensity for 177Lu-FF58 will be assessed and summarized using descriptive statistics. Dose intensity is computed as the ratio of actual cumulative dose received and actual duration of exposure.

SECONDARY OUTCOMES:
Overall response rate (ORR) | From start of study treatment until date of progression, assessed up to approximately 34 months
  ORR is defined as the proportion of patients with a BOR of complete response (CR) or partial response (PR) as per local review and according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 guidelines (non-GBM patients) or modified Response Assessment in Neuro- Oncology (mRANO) (GBM patients). It will be summarized along with the corresponding 90% exact CI using FAS.
Duration of Response (DOR) | From start of study treatment until date of progression, assessed up to approximately 34 months
  DOR is the time between the first documented response (CR or PR) and the date of progression as per local review and according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 guidelines (non-GBM patients) or modified Response Assessment in Neuro- Oncology (mRANO) (GBM patients), or death due to any cause. Here, death due to any cause is considered as an event to be conservative and align with PFS event definition. DOR may be presented graphically if enough events are available for analysis, using Kaplan Meier plots for all patients who achieved a CR/PR in the study. The median DOR and corresponding 90% CI will be presented. Analysis will include responders with confirmed responses.
Disease control rate (DCR) | From start of study treatment until date of progression, assessed up to approximately 34 months
  DCR is defined as the proportion of patients with a BOR of CR, PR, or stable disease as per local review and according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 guidelines (non-GBM patients) or modified Response Assessment in Neuro- Oncology (mRANO) (GBM patients). It will be summarized along with the corresponding 90% exact CI, using FAS.
Progression free survival (PFS) | From start of study treatment until date of progression, assessed up to approximately 34 months
  PFS is defined as the time from the date of start of treatment to the date of the first documented progression as per local review and according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 guidelines (non-GBM patients) or modified Response Assessment in Neuro- Oncology (mRANO) (GBM patients), or death due to any cause.
Area Under the Curve (AUC) from 177Lu-FF58 blood radioactivity data | Cycle 1 Day 1 (Pre-infusion, end of infusion, Post-dose (10 minutes(min), 30 min, 1 hours(hr), 2hr, 4hr, 6hr, 12hr)), Cycle 1 Day 2 (24hr), Cycle 1 Day 3 (48hr), Cycle 1 Day 4 (72hr), Cycle 1 Day 8 (168hr). Cycle=6 weeks or 3 weeks depending on schedule.
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity-based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. AUC from time zero to specified time point (mass x time x volume-1) will be listed and summarized using descriptive statistics.
Total body clearance from 177Lu-FF58 blood radioactivity data | Cycle 1 Day 1 (Pre-infusion, end of infusion, Post-dose (10 minutes(min), 30 min, 1 hours(hr), 2hr, 4hr, 6hr, 12hr)), Cycle 1 Day 2 (24hr), Cycle 1 Day 3 (48hr), Cycle 1 Day 4 (72hr), Cycle 1 Day 8 (168hr). Cycle=6 weeks or 3 weeks depending on schedule.
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. The total body clearance of drug from the plasma (volume x time-1) will be listed and summarized using descriptive statistics.
Observed maximum plasma concentration (Cmax) from 177Lu-FF58 blood radioactivity data | Cycle 1 Day 1 (Pre-infusion, end of infusion, Post-dose (10 minutes(min), 30 min, 1 hours(hr), 2hr, 4hr, 6hr, 12hr)), Cycle 1 Day 2 (24hr), Cycle 1 Day 3 (48hr), Cycle 1 Day 4 (72hr), Cycle 1 Day 8 (168hr). Cycle=6 weeks or 3 weeks depending on schedule.
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. Cmax will be listed and summarized using descriptive statistics.
Volume of distribution during the terminal phase following intravenous elimination (Vz) from 177Lu-FF58 blood radioactivity data | Cycle 1 Day 1 (Pre-infusion, end of infusion, Post-dose (10 minutes(min), 30 min, 1 hours(hr), 2hr, 4hr, 6hr, 12hr)), Cycle 1 Day 2 (24hr), Cycle 1 Day 3 (48hr), Cycle 1 Day 4 (72hr), Cycle 1 Day 8 (168hr). Cycle=6 weeks or 3 weeks depending on schedule.
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. Vz will be listed and summarized using descriptive statistics.
Terminal elimination half-life (T^1/2) from 177Lu-FF58 blood radioactivity data | Cycle 1 Day 1 (Pre-infusion, end of infusion, Post-dose (10 minutes(min), 30 min, 1 hours(hr), 2hr, 4hr, 6hr, 12hr)), Cycle 1 Day 2 (24hr), Cycle 1 Day 3 (48hr), Cycle 1 Day 4 (72hr), Cycle 1 Day 8 (168hr). Cycle=6 weeks or 3 weeks depending on schedule.
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. The half-life will be listed and summarized using descriptive statistics.
Urinary excretion of radioactivity expressed as a percentage of injected activity (%IA) | Cycle 1: Pre-infusion,beginning of infusion to first SPECT/CT image acquisition,first SPECT/CT image acquisition and 6 hours(hr) post-end-of infusion(EOI),6-24hr post-EOI,24-48hr post-EOI,48-72hr post-EOI. Cycle= 6 weeks or 3 weeks depending on schedule.
  Urine samples will be collected over specified time intervals and analysed for radioactivity. The radioactivity excreted in each interval as a percentage of injected activity (%IA) will be listed and summarized using descriptive statistics.
Time-activity curves (TACs) related to 177Lu-FF58 uptake in organs and tumor lesions | Cycle 1 Day 1, Cycle 1 Day 2 (24 hours (hr)), Cycle 1 Day 3 (48 hr), Cycle 1 Day 4 (72 hr), Cycle 1 Day 8 (168 hr). Cycle = 6 weeks or 3 weeks depending on schedule.
  Time-activity curves (TACs) for the various organs and tumor lesions will be produced as fraction of injected activity per gram of tissue (%IA/g) as a function of time.
Absorbed dose of 177Lu-FF58 | Cycle 1 Day 1, Cycle 1 Day 2 (24 hours (hr)), Cycle 1 Day 3 (48 hr), Cycle 1 Day 4 (72 hr), Cycle 1 Day 8 (168 hr). Cycle = 6 weeks or 3 weeks depending on schedule.
  The absorbed dose in target organs will be summarized with descriptive statistics. Lesion number will be assigned by dosimetry expert.
Incidence and severity of adverse events and serious adverse events of 68Ga-FF58 | From Imaging visit until 14 days after 68Ga-FF58 administration, or until first dose of study treatment
  The distribution of adverse events will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs) and Serious Adverse Event (TESAEs) due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.
Imaging properties: Visual and quantitative assessment (expressed as SUV) and tumor-to-background ratio (TBR) of 68Ga-FF58 uptake in organs and tumor lesions over time | From Imaging until 1 hour (hr), 2 hr and 3 hr after 68Ga-FF58 administration
  After 68Ga-FF58 administration, 68Ga-FF58 PET/CT or PET/MRI will be performed. The statistical analyses of imaging properties of 68Ga-FF58 will be descriptive in nature and will include summaries and graphical presentations of data. No formal testing will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- Novartis Investigative Site, Tel Aviv, Israel
- Novartis Investigative Site, Nijmegen, Netherlands
- Spain (2):
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CAAA604A12101 Clinical Trial Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18377
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=3008